CLINICAL TRIAL: NCT06156748
Title: CT Imaging for Guiding Postoperative Adjuvant Transarterial Chemoembolization for Hepatocellular Carcinoma
Brief Title: CT Imaging for Guiding PA-TACE for HCC
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Quan Xianyue, Academic Head of Department of Radiology, Zhujiang Hospital
Other Study IDs: 2019-KY-021-01
Record Dates: First submitted 2023-11-23; First posted 2023-12-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hepatectomy alone
  Interventions: Procedure: postoperative adjuvant transarterial chemoembolization
- PA-TACE

INTERVENTIONS:
Procedure: postoperative adjuvant transarterial chemoembolization — HCC patients received hepatectomy and PA-TACE.
  Groups: Hepatectomy alone

SUMMARY:
Postoperative adjuvant transarterial chemoembolization (PA-TACE) may improve survival outcomes in a subset of patients with resected hepatocellular carcinoma (HCC), reliable biomarkers for the criterion for the selection of candidates are lacking. The present study aimed to evaluate whether CT imaging can provide more value for predicting benefit from PA-TACE.

ELIGIBILITY:
Inclusion Criteria:

* CT scans acquired no more than one month before surgery
* Confirmation of HCC diagnosis by pathological examination
* Curative surgical resection

Exclusion Criteria:

* Prior antitumor treatment
* Macrovascular thrombosis or metastasis
* Perioperative mortality
* Unqualified image artifacts
* Tumor rupture
* MVI status not reported

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 1,488 patients (median age, 52 years [IQR, 45-61 years]; 1,309 male).
Sampling Method: Non-Probability Sample
Enrollment: 1770 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | the date of hepatectomy to the last follow-up or until death, whichever came first, assessed up to 120 months.
  Overall survival was calculated from the date of hepatectomy to the last follow-up or until death, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Liang X, Li Z, Liang J, Qi Z, Zhong L, Geng Z, Liang W, Quan X, Liang C, Liu Z. A novel stratification scheme combined with internal arteries in CT imaging for guiding postoperative adjuvant transarterial chemoembolization in hepatocellular carcinoma: a retrospective cohort study. Int J Surg. 2024 May 1;110(5):2556-2567. doi: 10.1097/JS9.0000000000001191. PMID 38377071